CLINICAL TRIAL: NCT04988568
Title: Experience of Patients Starting Hemodialysis: A Qualitative Study
Brief Title: Experience of Patients Starting Hemodialysis
Status: Completed | Type: Observational
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: SIH130
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None. This is a qualitative interview study. — There is no intervention in this study. This is a qualitative research study where patients will be interviewed.

SUMMARY:
Patients starting dialysis have significant and often daunting changes to their lifestyle, and investigators have only little information from the patient perspective on patient experiences during dialysis initiation. To explore patient perspectives when starting dialysis, this study aims to collect information on patient perspectives.

DETAILED DESCRIPTION:
Patients starting dialysis have significant and often daunting changes to their lifestyle, and investigators have only little information from the patient perspective on patient experiences during dialysis initiation. To explore patient perspectives when starting dialysis, this study aims to collect information on patient perspectives, understand what made patient experiences better, and what could further improve their experiences when patients first start dialysis. The investigators will enroll patients within 90 days of starting dialysis, and conduct semi-structured recorded interviews with patients. All patients will provide informed consent. The interviews will be transcribed verbatim.

* The transcripts will be reviewed line by line by qualitative researchers to identify concepts and themes, and will be developed into a coding schema.
* The preliminary themes will be discussed among the investigators to facilitate consensus.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving in-center hemodialysis care at Satellite Healthcare at the start of the study period.
* Patients who started with in-center hemodialysis as a first renal replacement therapy.
* Patients receiving dialysis for ≤ 90 days.

Exclusion Criteria:

* Age < 18 years.
* Unable to understand or communicate in English.
* Inability to participate because of cognitive impairment or active psychological condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All incident in-center hemodialysis patients meeting eligibility criteria at Satellite Healthcare, Inc., at IRB approved dialysis centers.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Experiences of patients starting dialysis. | One time interview.
  Collect information from interviews to understand the experiences of patients starting dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Wael F Hussein, MBBS, Principal Investigator — Satellite Healthcare, Inc.
Locations (17):
- United States (17):
  - Satellite Healthcare Los Gatos, Los Gatos, California
  - Satellite Healthcare Menlo Park, Menlo Park, California
  - Satellite Heathcare Milpitas, Milpitas, California
  - Satellite Dialysis Morgan Hill, Morgan Hill, California
  - Satellite Health Morgan Hill, Morgan Hill, California
  - Satellite Healthcare Mountain View, Mountain View, California
  - Satellite Healthcare Oakland, Oakland, California
  - Satellite Healthcare San Carlos, San Carlos, California
  - Satellite Healthcare East San Jose, San Jose, California
  - Satellite Health Blossom Valley, San Jose, California
  - Satellite Health San Teresa, San Jose, California
  - Satellite Healthcare SIlver Creek, San Jose, California
  - Satellite Health South San Jose, San Jose, California
  - Satellite Healthcare Evergreen, San Jose, California
  - Satellite Dialysis San Leandro, San Leandro, California
  - Satellite Healthcare West San Leandro, San Leandro, California
  - Satellite Dialysis San Mateo, San Mateo, California

IPD SHARING:
Plan to Share IPD: No
No individual person data will be available to anyone other than Satellite Healthcare Research employees.